CLINICAL TRIAL: NCT00188643
Title: Double-Blind, Acute Depression Study Comparing Venlafaxine XR and Lamotrigine When Added to Mood Stabilizer in the Treatment of Bipolar Depression
Brief Title: Venlafaxine Versus Lamotrigine in the Treatment of Bipolar I/II Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2005-02

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder, Depression, Anticonvulsants, Antidepressants
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Venlafaxine Hydrochloride; Lamotrigine

INTERVENTIONS:
Drug: Venlafaxine and Lamotrigine

SUMMARY:
The primary objective of this study is to assess the efficacy of venlafaxine XR and lamotrigine when each is added to mood stabilizer therapy in patients with acute depressive episodes of bipolar I or Bipolar II disorder. Efficacy of therapy will be evaluated using improvements in clinical symptomatology after 8 weeks of treatment as measured by reductions on the Hamilton Depression Rating Scale (HDRS-29) total score >50% from baseline. We also would like to assess the efficacy of venlafaxine XR and lamotrigine when each is added to mood stabilizer therapy in improving clinical symptomatology after 8 weeks of therapy as well as to evaluate the side effect profile, safety and tolerability of venlafaxine XR and lamotrigine.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the efficacy of venlafaxine XR and lamotrigine when each is added to mood stabilizer therapy in patients with acute depressive episodes of bipolar I or Bipolar II disorder. Efficacy of therapy will be evaluated using improvements in clinical symptomatology after 8 weeks of treatment as measured by reductions on the Hamilton Depression Rating Scale (HDRS-29) total score >50% from baseline. We also would like to assess the efficacy of venlafaxine XR and lamotrigine when each is added to mood stabilizer therapy in improving clinical symptomatology after 8 weeks of therapy as well as to evaluate the side effect profile, safety and tolerability of venlafaxine XR and lamotrigine.

ELIGIBILITY:
Inclusion Criteria:

* 1. Meets DSM-IV criteria for a diagnosis of Bipolar I disorder, most recent episode depression, or bipolar II disorder, most recent episode depression using the structured clinical interview for DSM-IV Axis 1 disorders 2. Subjects must have a Hamilton depression rating scale score of >16. 3. Patients at visit 1 must have documented trials (levels must be obtained) of their mood stabilizer for at least 2 weeks 4. Subjects must be between the ages of 18-70, male or female 5. Treatment with oral antipsychotics, anticonvulsants or benzodiazepines prior to enrolment or during the study will be permitted, but not other antidepressants.

  6. Female patients of childbearing potential must be using a medically accepted means of contraception.

  7. Patient is judged by the investigator to be in generally good health 8. Education level and a degree of understanding is such that the patient can communicate effectively with the investigator.

  9. Patient must be capable of providing informed consent.

Exclusion Criteria:

* 1. Treatment with antidepressant medication within one day prior to visit 1 or during the protocol.

  2. Patients previously showing poor therapeutic response to venlafaxine XR or lamotrigine 3. Judged clinically to be at serious suicidal risk. 4. DSM-IV criteria for substance dependence (except nicotine or caffeine) within the past 30 days 5. Course of ECT (electroconvulsive therapy) in the preceding 4 weeks prior to visit 1 or during the protocol.

  6. Patients who suffer from a major neurological or medical illness. 7. Current diagnosis of schizophrenia or other psychotic disorders as defined in the DSM-IV 8. Uncorrected hypothyroidism or hyperthyroidism 9. Female patients who are either pregnant or nursing 10. Elevated thyroid stimulating hormone (TSH).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-01; Study Completion 2007-01

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale, 21 item

SECONDARY OUTCOMES:
Young Mania Rating Scale (YMRS)
Montgomery Asberg Depression Rating Scale (MADRS)
Clinical Global Impression (CGI-I, CGI-S)
Quality of Life Enjoyment
Global Assessment of Functioning

CONTACTS AND LOCATIONS:
Overall Officials: Roger McIntyre, MD,FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada